CLINICAL TRIAL: NCT06521892
Title: The Effect of Social Surveillance and Health Education Interventions Non-prescription Dispensing of Antibiotics in Community Pharmacies: a Randomized Controlled Trial
Brief Title: Interventions on Non-prescription Dispensing of Antibiotics in Community Pharmacies
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoxv Yin, PhD, Professor and Head of Social Medicne and Health Management Department, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HuazhongU20240720
Record Dates: First submitted 2024-07-20; First posted 2024-07-26 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Non-Prescription Drug Misuse; Acute Respiratory Tract Infection
Keywords: antibiotic; community pharmacy; non-prescription; randomized controlled trial
MeSH Terms: conditions — Drug Misuse

STUDY DESIGN:
Intervention Model Description: In parallel arm design, subjects are randomized to one or more study arms and each study arm will be allocated a different intervention. After randomization each subject stays in their assigned treatment arm for the duration of the study. Subjects receive the same treatment throughout the trial. The results are then compared
Who Masked: Participant, Investigator
Masking Description: Pharmacies participating in the study did not know which group they were assigned to. Standardized patient surveyors also did not know which group of pharmacies they surveyed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants in intervention group will receive social supervision and health education interventions.
  Interventions: Behavioral: social surveillance and health education interventions
- control group (No Intervention): Participants in control group will receive routine drug supervision and management measures.

INTERVENTIONS:
Behavioral: social surveillance and health education interventions — Social surveillance: In the intervention group retail pharmacies posted or hung signs "antibiotics need to be purchased by prescription, if found without prescription sales, welcome to call 12315 hotline to report", to form social supervision intervention.
  Health education: On-site training for retail pharmacy staff, inviting respiratory physicians and pediatricians to give health education lectures on disease diagnosis, treatment and medication.
  Arms: intervention group

SUMMARY:
This study was a randomized controlled trial conducted in community pharmacies. Empirical data were collected primarily using standardized patient methods. In Hubei Province, 400 community pharmacies were randomly selected and assigned to the intervention group and the control group according to the ratio of 1:1. A one-month intervention was conducted in community pharmacies in the intervention group, which included both social surveillance and health education. First, on-site training was provided to community pharmacy staff. Respiratory physicians and pediatricians were invited to give health education lectures on disease diagnosis and treatment, medication use, etc. Second, signs were posted or hung in the community pharmacies of the intervention group, saying that "antibiotics need to be purchased with a prescription, and you are welcome to call the 12315 hotline to report if you find any sales without a prescription", in order to open up the channels of social supervision and to form a social surveillance intervention. The control group only received the regular drug supervision and management measures in Hubei Province. The primary outcome is to observe the proportion of community pharmacies selling antibiotics without a prescription.

ELIGIBILITY:
Inclusion Criteria:

* The qualification of retail pharmacies to sell antimicrobial drugs complies with relevant regulations and requirements, ensuring that the study participants operate legally within the regulatory framework.
* Pharmacies located in Hubei Province.

Exclusion Criteria:

* The retail pharmacy plans to undergo major changes during the study period, such as relocation, renovation, shutdown, or closure;
* Retail pharmacies that refused to respond to the call for training from the Hubei Provincial Drug Administration;
* Participants had poor compliance and do not participate in the intervention as required by the trial on multiple occasions;
* Subjects withdrew from the study on their own or were lost to follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of antibiotics dispensing without a prescription | baseline, First month after intervention, 3, 6, and 12 months after intervention
  Proportion of antibiotics dispensing without a prescription measured by standardized patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Provincial Drug Administration, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No